CLINICAL TRIAL: NCT01546051
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetic and Food Effect of BCI-838; and, An Open-Label Minidose Bioavailability Study to Compare Several BCI-632 Pro-drug Candidates in Healthy Male Subjects
Brief Title: A Study of BCI-838 and Several BCI-632 Prodrugs in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrainCells Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BCI-632-CL-002
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: metabotropic glutamate receptors 2 and 3; antagonist; mGluR; ketamine; BDNF; Depression; Major Depressive Disorder; Mood Disorder; Treatment Resistant Depression; Phase 1 safety, tolerability and pharmacokinetics study
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Mood Disorders; Depressive Disorder, Treatment-Resistant | interventions — BCI-838

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BCI-838 Food Effect Dosing Arm 1 (Experimental): Eight subjects will be enrolled, 6 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838
- BCI-838 Fasted Dosing (100 & 300 mg) (Experimental): Eight subjects will be enrolled, 6 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838
- BCI-1038, BCI-1206 & BCI-1283 (Experimental): Six subjects will be enrolled, all 6 will receive single doses of BCI-1038, BCI-1206 and BCI-1283.
  Interventions: Drug: BCI-1038, BCI-1206 & BCI-1283
- BCI-838 Fasted Dosing (900 mg) (Experimental): Eight subjects will be enrolled, 6 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838

INTERVENTIONS:
Drug: BCI-838 — BCI-838 100 mg and 300 mg or matching placebo administered as single oral doses under fasted conditions in a sequential design
  Arms: BCI-838 Fasted Dosing (100 & 300 mg)
Drug: BCI-838 — BCI-838 administered as a single 30 mg oral dose or matching placebo under fasted and fed conditions in a crossover design
  Arms: BCI-838 Food Effect Dosing Arm 1
Drug: BCI-1038, BCI-1206 & BCI-1283 — Three new pro-drugs administered as a 1 mg single oral doses under fasted conditions in a sequential design
  Arms: BCI-1038, BCI-1206 & BCI-1283
Drug: BCI-838 — BCI-838 900 mg or matching placebo administered as a single oral dose under fasted conditions
  Arms: BCI-838 Fasted Dosing (900 mg)

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of BCI-838, its metabolite BCI-632 and several new pro-drugs in healthy male subjects.

DETAILED DESCRIPTION:
The first phase of this study will evaluate the safety and tolerability of BCI-838 following oral administration of single doses of BCI-838 in healthy male subjects. The pharmacokinetics of BCI-838 and its metabolite BCI-632 following single ascending doses of BCI-838 will be evaluated, as will the effect of food on the pharmacokinetics of BCI-838 and its metabolite following single oral doses of BCI-838 in healthy male subjects.

The second phase of this study will evaluate and compare the relative bioavailability and PK of the metabolite BCI-632 following single oral administration of several new pro-drug candidates in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult male healthy volunteer, 18-55 years of age
* Body Mass Index (BMI) between 18.0 to 30.0 kg/m2 inclusive
* Good general health as determined by medical history and physical examination with no clinically significant medical findings and no clinically relevant medical or surgical history and no acute or ongoing conditions within the past 30 days
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Clinically significant medical abnormality, chronic disease or history or presence of significant pulmonary, gastrointestinal, metabolic, cardiac, hepatic, renal or neurological disorder
* History or current use of alcohol abuse or drug addiction
* Participation in a drug study within 60 days prior to drug administration.
* Participation in more than 3 other drug studies in the 10 months preceding the start of this study
* Donation or blood loss of more than 50 mL of blood within 60 days prior to the first drug administration. Donation of more than 1.5 liters of blood in the 10 months preceding the start of this study
* Illness within 5 days prior to drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety | 7 days
  Safety will be evaluated by adverse events, vital signs, ECG, clinical labs, and physical exam.

SECONDARY OUTCOMES:
Cmax, tmax, t1/2 , AUC, CL/F, Vz/F, and Kel of BCI-838 and BCI-632 | predose and at specified intervals up to 72 hours post-dose
  The pharmacokinetics of BCI-838 and its metabolite BCI-632, an assessment of the dose proportionality of the pharmacokinetics following single ascending doses of BCI-838, and an evaluation of the relative bioavailability and pharmacokinetics of the metabolite BCI-632 following oral administration of several new pro-drug candidates will be completed by assessment of Cmax, tmax, t1/2 , AUC, CL/F, Vz/F, and Kel.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International, Zuidlaren, Netherlands